CLINICAL TRIAL: NCT00353210
Title: The Derivation of Human Embryonic Stem Cell Lines From PGD Embryos
Status: Recruiting | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: 24-23.04.04-HMO-CTIL
Record Dates: First submitted 2006-07-16; First posted 2006-07-18 (Estimated); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Infertility
Keywords: IVF; embryos; research; donation; surplus; stem cells; abnormal embryo; screening
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — PGD embryos derived from IVF that are determined to be not suitable for return to the uterus of the female due to the results of PGD analysis and only then the parents decide to donate them to our program for use in hESC research.
Oversight: Data Monitoring Committee: No

SUMMARY:
Human embryonic stem cells (hESCs) are isolated from the early human embryo and have the capability to proliferate indefinitely in culture and to develop into nearly every cell of the human body. hESC are important for studying developmental biology and for cell replacement therapies for the treatment of degenerative human diseases. An additional use for embryonic stem cells would be for the in vitro study of diseases. hESC lines derived from embryos diagnosed as abnormal by PGD testing would afford such models for study. Because embryos tested by PGD and found to be abnormal would only under rare circumstances be transferred to the uterus of a woman (and in most cases would be discarded), the derivation of new hESC lines from these embryos would provide a viable less ethically-objectionable source of cells with which to study the mechanisms of differentiation and developmental biology.

DETAILED DESCRIPTION:
Embryonic stem cells are pluripotent cells that are derived from the early stage embryo (the blastocyst stage). Embryonic stem cells are the only cells that have the ability to provide an unlimited source of daughter cells and can differentiate into virtually any cell of the body.

Human embryonic stem cell lines have previously been derived from supernumerary embryos donated by couples undergoing IVF treatment. Thomson was the second in the world to isolate human embryonic stem cells. We derived six human embryonic stem cell lines, which are registered with the National Institute of Health and are eligible for American federal funding for research. We are widely distributing our cell lines to many researchers worldwide.

The key features of human embryonic stem cells are their potential of unlimited proliferation in culture, and their ability to differentiate into a large variety of somatic cells of the body. Our group was the first to show this capability in culture (1). Our results, and the results of other groups show that human embryonic stem cells can differentiate in culture into nerve cells, blood cells, pancreatic cells that secrete insulin, heart muscle cells, and others. Given the key properties of human embryonic stem cells, they are expected to have far reaching applications in basic scientific research, development of new drugs, and may serve as an unlimited donor source of cells for transplantation.

Embryonic stem cells will be recovered from human blastocysts donated to stem cell research by couples that have undergone preimplantation genetic diagnosis (PGD) of their embryos during IVF. In PGD, a number of embryos are generated by routine IVF, and cellular material is then taken as a biopsy from early human embryos that have been cultured in vitro. Embryos that are found to be genetically normal are selectively transferred to the uterus. A portion of the tested embryos will not have a diagnosis or will be found to contain specific genetic mutations or chromosomal aberrations. After discussion with the couple and subjected to their consent, these embryos will not be implanted in the potential mother for the purposes of pregnancy. It should be noted that in cases of uncertain diagnosis the couples may elect to transfer the embryos and perform prenatal diagnosis and pregnancy termination in cases where the fetus is found to be affected. Otherwise, the affected embryos or those without a certain diagnosis are truly surplus embryos that are routinely discarded. We wish to derive human embryonic stem cell lines from these embryos, since they will contain a specific mutation or chromosomal aberration that will be of interest to the research community. The genetically abnormal stem cells, that will be derived from these PGD-tested embryos, will be useful tools for the investigation of early development, cell function, disease progression, and for the efficacy or toxicity of drug therapies for the genetic abnormalities that they will carry. Derivation of human ES cell lines that harbor a specific gene defect will have great importance in the study and development of treatments for certain inheritable disorders. In addition, they may be employed for the development of gene therapy strategies designed for potential treatment of specific inherited disorders.

It should be stressed that the embryos that will be recruited for this study would have been discarded in any event, and would not have been implanted to produce a child. The embryos, while precious, will contain or will be suspected to contain undesired chromosomal or single gene defects, and will not have been deemed acceptable for transfer by the couple undergoing IVF. By contrast, these embryos, while not suitable for the purposes of producing healthy offspring, are valuable to stem cell research as key tools for the study of specific human disorders, therapies, for the investigation of early human development, in the derivation of new medications to treat diseases, and possibly to correct genetic defects. Rather than simply discarding and destroying the stem cells within these faulty embryos, they will be salvaged and utilized in the derivation of new disease-specific human embryonic stem cell lines.

Since the new lines derived from PGD embryos will be utilized for research purposes only, the derivation of new embryonic stem cell lines will occur under GLP conditions, utilizing predetermined acceptable raw materials and methods. These lines may be characterized and safety tested like the non-PGD-tested lines after manufacturing in the Research and Development Laboratory of the Goldyne Savad Institute of Gene Therapy.

The PGD-tested embryos will be obtained under full informed consent prior to their utilization in research. Voluntary donations of embryos will be recruited, in accordance with existing regulations and legislation. The donors will be approached only after the decision to discard the genetically abnormal embryos has been independently made. IVF staff will approach the donors, answer any questions they may have, and obtain their permission prior to utilization of their embryos. Because of the many ethical concerns regarding the removal of fetal cells from human embryos, we are extremely sensitive to the moral debates as to the "rights" and the "personage" of an embryo. Once obtained, the embryos will be developed to the blastocyst stage and the stem cells removed, according to accepted protocols for human embryonic stem cell line development. No identifiable features of the donor couple, exclusive of the known genetic mutation, will be attached to any of the embryos donated to research.

ELIGIBILITY:
Inclusion Criteria:

* Couple has derived embryos by IVF.
* Couple has tested these embryos by PGD and does not want to utilize the embryos to build their families.
* Couple signs informed consent.

Exclusion Criteria:

* Couple does not sign informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Embryo donors of embryos that have undergone PGD analysis after IVF which the donors have no intention of using for family-building purposes.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2004-04-06 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin E. Reubinoff, M.D. PhD., Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Background] Pickering SJ, Braude PR, Patel M, Burns CJ, Trussler J, Bolton V, Minger S. Preimplantation genetic diagnosis as a novel source of embryos for stem cell research. Reprod Biomed Online. 2003 Oct;7(3):353-64. doi: 10.1016/s1472-6483(10)61877-9. PMID 14653899
- See also: website about the Hadassah hESC Research Center clinical-grade cell lines — https://hhesc.co.il